CLINICAL TRIAL: NCT05918367
Title: Multicenter Ventral Mesh Rectopexy Registry Collaborative
Acronym: M2R2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 001130
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-06

CONDITIONS: Pelvic Organ Prolapse; Rectocele; Enterocele; Rectal Prolapse; Descending Perineum Syndrome; Surgery
Keywords: Posterior pelvic organ prolapse; descending perineum; ventral mesh rectopexy; functional outcome
MeSH Terms: conditions — Pelvic Organ Prolapse; Rectocele; Hernia; Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter observational study is to collect data prospectively of patients with pelvic organ prolapse undergoing ventral mesh rectopexy (as well as rectoceles, entero-/sigmoidoceles/ intussusception/ rectal prolapse or combined) by laparoscopy or robotic surgery and to evaluate the longterm functional outcomes.

Secondly complications (mesh erosions, recurrence, reoperations) are evaluated.

Following main questions will be analysed - other can follow in consultation with the collaborative

1. Is VMR the technique of choice for treatment of rectoceles? Functional results - recurrence - mesh related complications
2. Has a perineal descent an impact on the functional outcome of ventral mesh rectopexy perfored for external rectal prolaps, internal rectal prolaps, rectocele, enterocele, sigmoidcele or combined pelvic organ prolapse?

DETAILED DESCRIPTION:
The study M2R2 is a multicentre registry based on the still ungoing monocentre study in the University Hospital of Antwerp.

Pelvic organ prolapse (POP) is a benign condition in which pelvic organs prolapse beyond their normal anatomical position due to weakening or damage to the pelvic floor muscles and other supporting tissues.[1] The incidence increases with age, multiparity, vaginal delivery and obesity.[2] POP can cause urinary, sexual and bowel complaints with a huge impact on quality of life.[3,4] Patients with posterior compartment prolapse may include symptoms of vaginal swelling, heaviness, perineal pressure and/or obstructive defecation with fragmented stools, need for hard straining, feeling of incomplete emptying, splinting, faecal urgency and even incontinence.[4] Ventral mesh rectopexy is surgical technique used to treat posterior compartment prolapse (rectocele, enterocele, sigmoidocele, rectal prolapse, combination) in patients with symptoms where conservative therapy fails or is ineffective. In this procedure, a mesh is placed between the back wall of the vagina and the rectum, the rectovaginal septum. This is attached at the level of the bone higher up (the promontorium) so that the back wall of the vagina is reinforced, preventing the prolapse to recurre.This technique was first described as technique to treat rectal prolapse by d'Hoore, a colorectal surgeon and widely accepted given the feasible transabdominal technique with good functional results. However, whether this technique gives also effective long-term anatomical and functional outcomes for rectoceles, enteroceles/sigmoidoceles +/- perineal descent, besides rectal prolapse, is not known.[5,6] Sometimes a combined procedure is necessary in which the anterior compartment (bladder) and/or middle compartment (cervix/vagina tip) is also reinforced.

The main objective of this registry is to collect data prospectively of patients with pelvic organ prolapse undergoing ventral mesh rectopexy (as well as rectoceles, entero-/sigmoidoceles/ intussusception/ rectal prolapse or combined) by laparoscopy or robotic surgery and to evaluate the longterm functional outcomes.

Secondly complications (mesh erosions, recurrence, reoperations) are evaluated.

The patients will be recruited from outpatient clinic of abdominal surgery in the participating centers. The treating physician recruits patients.

Methods and analysis

1. Data registry Parameters will be registered by means of case record form: History of the patient, urinary, prolapse, defecatory complaints, MRI or CR CCD if performed, anal manometry if performed, results of pelvic floor physiotherapy if performed. Surgical technique, operation time/length of stay and complications.
2. Questionnaire send to the patients at 5 time points

   Preoperative - 3 months - 1 year - 3 years - 5 years postoperative

   Questionnaires consisting of different topics I. In female: questions about childbirth (only preoperative) II. Medication III. Inventarisation of pelvic floor (dys)- function: PFDI-20 IV. Intestinal function and constipation
   * Wexner Vaizey-score
   * Low anterior resection syndrome score (LARS)
   * Bristol stool chart
   * Rome IV criteria functionam obstipation
   * Rome IV criteria IBS
   * CCS (Wexner constipation score)

   V. Urinary (ICIQ-SF) VI. Seksuality (PISC-IR) VII. Impact of pelvic floor problem on quality of life (PISQ-7) VIII. Subjective satisfaction after surgery
3. Data management

Collected data will be entered in a case record form by the treating physician of the participating centre or by assigned study staff using the RedCap platform. Patients will be coded to insure patient anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of posterior pelvic organ prolaps planned for laparoscopie or robotic ventral mesh rectopexy with or without concomittant surgery.
* All patients 18 years or older and are able to complete a written informed conscent are eligble for inclusion.

Exclusion Criteria:

1. Inability to complete a written informed conscent
2. Pregnant women
3. No email adress available to send the questionnaires to
4. Language barrier or impossiblity to fill in the questionnaires (at the discretion oft he treating physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pelvic organ prolapse undergoing ventral mesh rectopexy (as well as rectoceles, entero-/sigmoidoceles/ intussusception/ rectal prolapse or combined)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 5 years
  Evaluation of the long-term functional outcomes of ventral mesh rectopexy (VMR) for posterior organ prolapse. Is VMR the surgical technique of choice for treatment of rectoceles?
Has perineal descent has an impact on the functional outcome of ventral mesh rectopexy performed for external rectal prolaps, internal rectal prolaps, rectocele, enterocele, sigmoidocele or combined pelvic organ prolapse? | 5 years

SECONDARY OUTCOMES:
recurrence of posterior pelvic organ prolapse - new onset of symptoms | 5 years
mesh related complications | 5 years

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - UZ Brussel, Brussels
  - University Hospital Antwerp, Edegem
  - AZ Jan Palfijn, Ghent
  - Jessa ziekenhuis, Hasselt
  - AZ Delta Roeselare, Roeselare

REFERENCES:
- [Result] Weintraub AY, Glinter H, Marcus-Braun N. Narrative review of the epidemiology, diagnosis and pathophysiology of pelvic organ prolapse. Int Braz J Urol. 2020 Jan-Feb;46(1):5-14. doi: 10.1590/S1677-5538.IBJU.2018.0581. PMID 31851453
- [Result] Vergeldt TF, Weemhoff M, IntHout J, Kluivers KB. Risk factors for pelvic organ prolapse and its recurrence: a systematic review. Int Urogynecol J. 2015 Nov;26(11):1559-73. doi: 10.1007/s00192-015-2695-8. Epub 2015 May 13. PMID 25966804
- [Result] Pelvic Organ Prolapse: ACOG Practice Bulletin, Number 214. Obstet Gynecol. 2019 Nov;134(5):e126-e142. doi: 10.1097/AOG.0000000000003519. PMID 31651832
- [Result] Doumouchtsis SK, Raheem AA, Milhem Haddad J, Betschart C, Contreras Ortiz O, Nygaard CC, Medina CA, La Torre F, Iancu G, Cervigni M, Zanni G. An update of a former FIGO Working Group Report on Management of Posterior Compartment Prolapse. Int J Gynaecol Obstet. 2020 Feb;148(2):135-144. doi: 10.1002/ijgo.13006. Epub 2019 Nov 19. PMID 31628853
- [Result] D'Hoore A, Penninckx F. Laparoscopic ventral recto(colpo)pexy for rectal prolapse: surgical technique and outcome for 109 patients. Surg Endosc. 2006 Dec;20(12):1919-23. doi: 10.1007/s00464-005-0485-y. PMID 17031741
- [Result] D'Hoore A, Cadoni R, Penninckx F. Long-term outcome of laparoscopic ventral rectopexy for total rectal prolapse. Br J Surg. 2004 Nov;91(11):1500-5. doi: 10.1002/bjs.4779. PMID 15499644